CLINICAL TRIAL: NCT00084513
Title: Phase I of Trastuzumab and Imatinib Mesylate (Gleevec®, Formerly Known as STI-571) in Patients With Recurrent or Metastatic Her-2/Neu Expressing Cancer
Brief Title: Trastuzumab and Imatinib Mesylate in Treating Patients With Recurrent or Metastatic HER2/Neu-Expressing Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000365451; P30CA006927 (NIH); FCCC-03041; NOVARTIS-FCCC-03041
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Trastuzumab; Imatinib Mesylate

INTERVENTIONS:
Biological: trastuzumab
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth and by stopping blood flow to the tumor. Giving trastuzumab together with imatinib mesylate may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib mesylate when given together with trastuzumab in treating patients with recurrent or metastatic HER2/neu-expressing (producing) cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of imatinib mesylate when administered with trastuzumab (Herceptin®) in patients with recurrent or metastatic HER2/neu-overexpressing cancer.
* Determine response in patients treated with this regimen.

Secondary

* Correlate the number of circulating tumor cells with radiographic imaging in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of imatinib mesylate.

Patients receive trastuzumab (Herceptin®) IV over 90 minutes on day 1 and oral imatinib mesylate once or twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 9-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed cancer that overexpresses HER2/neu, measured 3+ by immunohistochemistry or positive by fluorescence in situ hybridization

  * Recurrent or metastatic disease
* Meets 1 of the following criteria for measurable or evaluable disease:

  * Unidimensionally measurable disease at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Evaluable disease, defined as a lesion on physical examination or imaging study that can be assessed as to changes in size but cannot be clearly measured in 1 dimension (e.g., pleural effusions, ascites, or bone disease)
* No carcinomatous meningitis or untreated/uncontrolled metastatic brain parenchymal disease

  * Prior controlled brain parenchymal disease allowed provided at least 8 weeks since prior therapy AND no symptomatic progression off corticosteroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* ALT and AST ≤ 2.0 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.0 times ULN
* Bilirubin ≤ 1.3 mg/dL
* No known chronic liver disease (i.e., chronic active hepatitis or cirrhosis)

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* Ejection fraction ≥ lower limit of normal by MUGA
* No uncontrolled or significant cardiovascular disease
* No myocardial infarction within the past 6 months
* No ischemic heart disease requiring medication
* No congestive heart failure

Pulmonary

* No uncontrolled or significant pulmonary disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No active unresolved infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior trastuzumab (Herceptin®) allowed
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF) to support blood counts
* No other concurrent anticancer biologic agents

Chemotherapy

* Prior chemotherapy for metastatic disease allowed
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent anticancer chemotherapy

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* More than 2 weeks since prior major surgery

Other

* At least 7 days since prior antibiotics
* No concurrent parenteral antibiotics
* No other concurrent anticancer agents
* No other concurrent investigational drugs
* No concurrent therapeutic anticoagulation with warfarin

  * Concurrent mini-dose warfarin (1 mg/day) for prophylaxis of central venous catheter thrombosis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2004-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of imatinib mesylate given concurrently with trastuzumab (Herceptin®) as measured by CTC v 3.0 at course 1
Response as measured by RECIST criteria every 9 weeks

SECONDARY OUTCOMES:
Circulating tumor cells in blood as measured by Immunicom Cell PrepTM at baseline, every 3 weeks until week 9, and then with each disease re-evaluation
Phosphorylation status of AKT, extracellular signal-regulated kinase (ERK), and KIT as measured by western blot and/or immunohistochemistry at baseline and week 9

CONTACTS AND LOCATIONS:
Overall Officials: Margaret von Mehren, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States